CLINICAL TRIAL: NCT01882465
Title: Corneal Staining Associated With Daily Disposable Beauty Contact Lenses
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Johnson & Johnson Vision Care, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: CR-5360
Record Dates: First submitted 2013-06-07; First posted 2013-06-20 (Estimated); Results first posted 2016-10-05 (Estimated); Last update posted 2018-06-19 (Actual); Status verified 2016-11

CONDITIONS: Refractive Error
MeSH Terms: conditions — Refractive Errors

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (6):
- etafilcon A/2-HEMA, EGDMA/hefilcon A (Other): Subjects were randomized to one of six unique sequences. Subjects randomized to this sequence will wear the etafilcon A lens first, the 2-HEMA, EGDMA Non-ionic material lens second and the hefilcon A lens third. The lenses are to be worn in a daily wear modality, and disposed of at the end of each follow-up visit.
  Interventions: Device: etafilcon A; Device: 2-HEMA, EGDMA Non-ionic; Device: hefilcon A
- etafilcon A/hefilcon A/2-HEMA, EGDMA Non-ionic (Other): Subjects were randomized to one of six unique sequences. Subjects randomized to this sequence will wear the etafilcon A lens first, the hefilcon A lens second and the 2-HEMA, EGDMA Non-ionic material lens third. The lenses are to be worn in a daily wear modality, and disposed of at the end of each follow-up visit.
  Interventions: Device: etafilcon A; Device: 2-HEMA, EGDMA Non-ionic; Device: hefilcon A
- 2-HEMA, EGDMA Non-ionic/etafilcon A/hefilcon A (Other): Subjects were randomized to one of six unique sequences. Subjects randomized to this sequence will wear the 2-HEMA, EGDMA Non-ionic material lens first, the etafilcon A lens second and the hefilcon A lens third. The lenses are to be worn in a daily wear modality, and disposed of at the end of each follow-up visit.
  Interventions: Device: etafilcon A; Device: 2-HEMA, EGDMA Non-ionic; Device: hefilcon A
- 2-HEMA, EGDMA Non-ionic/hefilcon A/etafilcon A (Other): Subjects were randomized to one of six unique sequences. Subjects randomized to this sequence will wear the 2-HEMA, EGDMA Non-ionic material lens first, the hefilcon A lens second and the etafilcon A lens third. The lenses are to be worn in a daily wear modality, and disposed of at the end of each follow-up visit.
  Interventions: Device: etafilcon A; Device: 2-HEMA, EGDMA Non-ionic; Device: hefilcon A
- hefilcon A/2-HEMA, EGDMA Non-ionic/etafilcon A (Other): Subjects were randomized to one of six unique sequences. Subjects randomized to this sequence will wear the hefilcon A lens first, the 2-HEMA, EGDMA Non-ionic material lens second and the etafilcon A lens third. The lenses are to be worn in a daily wear modality, and disposed of at the end of each follow-up visit.
  Interventions: Device: etafilcon A; Device: 2-HEMA, EGDMA Non-ionic; Device: hefilcon A
- hefilcon A/etafilcon A /2-HEMA, EGDMA Non-ionic (Other): Subjects were randomized to one of six unique sequences. Subjects randomized to this sequence will wear the hefilcon A lens first, the etafilcon A lens second and the 2-HEMA, EGDMA Non-ionic material lens third. The lenses are to be worn in a daily wear modality, and disposed of at the end of each follow-up visit.
  Interventions: Device: etafilcon A; Device: 2-HEMA, EGDMA Non-ionic; Device: hefilcon A

INTERVENTIONS:
Device: etafilcon A — Lenses to be worn in a daily wear modality, and disposed of at the end of each follow-up visit.
  Other Names: 1-Day Acuvue DEFINE (Vivid)
Device: 2-HEMA, EGDMA Non-ionic — Lenses to be worn in a daily wear modality, and disposed of at the end of each follow-up visit.
  Other Names: SEED Eye Coffret 1-Day UV Rich Make
Device: hefilcon A — Lenses to be worn in a daily wear modality, and disposed of at the end of each follow-up visit.
  Other Names: Ticon Cosmetic Daily Black

SUMMARY:
Limbal ring contact lenses enhance the look of the eye by adding pigmentation in a ring pattern to the contact lens. The purpose of this investigation is to determine if corneal staining increase is dependent upon the lens pigment location.

ELIGIBILITY:
Inclusion Criteria:

1. The subject must read, understand, and sign the STATEMENT OF INFORMED CONSENT and receive a fully executed copy of the form.
2. Fluency in English and ability to read and understand written English.
3. The subject must be able and willing to adhere to the instructions set forth in this clinical protocol.
4. The subject must be between 18 and 35 years of age.
5. The subject must be an adapted (minimum of 4 week history of daily wear prior to the baseline study visit) soft contact lens wearer in both eyes.
6. The subject must be East or Southeast Asia descent, e.g. ethnic Chinese, Japanese, Korean, Malay, Vietnamese, Indonesian, Filipino, etc. by self-report.
7. The subject must come in with a current (no more than 12 month old) spectacle or contact lens prescription as indicated. (NB: Emmetropic subjects who wear contact lenses for enhancement purposes only will also require a current contact lens prescription).
8. The subject's vertex corrected spherical equivalent distance refraction must be in the range of PLANO to -6.00 Diopter (D) in each eye.
9. The subject must have best corrected visual acuity on +0.24 logMAR (equivalent to 20/30 (-2)) or better in each eye.
10. The subject must own a wearable pair of spectacles (as indicated by current prescription) and wear them to all visits including the screening visit as required for vision correction. They must be willing to wear their spectacles during the 24 hour washout period leading up to each treatment visit (NB: Emmetropic subjects who do not own spectacles must agree to no lens wear on all visit days including the screening visit).
11. The subject must have normal eye (i.e., no ocular medications or infections of any type).

Exclusion Criteria:

1. Are currently pregnant or lactating, determined by self-report (subjects who become pregnant during the study will be discontinued).
2. Have any ocular or systemic allergies or diseases that may interfere with contact lens wear.
3. Have any systemic disease, autoimmune disease, or use of medication, which may interfere with contact lens wear. This may include, but may not be limited to diabetes, hyperthyroidism, recurrent herpes simplex/zoster, Sjogren's syndromes, xerophthalmia, acne rosacea, Stevens-Johnson syndromes.
4. Use any topical medication such as eye drops or ointment.
5. Have entropion, ectropion, extrusions, chalazia, recurrent styes, glaucoma, history of recurrent corneal erosions, or aphakia.
6. Had any previous, or have planned, ocular or intraocular surgery (e.g., cataract surgery, radial keratotomy, photorefractive keratectomy (PRK), laser-assisted in situ keratomileusis (LASIK).
7. Have any grade 3.0 or greater slit lamp findings (e.g., edema, corneal neovascularization, corneal staining, tarsal abnormalities, conjunctival injection) on the Efron classification scale or any other ocular abnormality that may contraindicate contact lens wear.
8. Have any known hypersensitivity or allergic reaction to contact lenses (as assessed by ocular history).
9. Have any ocular infection.
10. Have any corneal distortion resulting from previous hard or rigid gas permeable contact lens wear.
11. Have participated in any contact lens or lens care product clinical trial within 14 days prior to study enrollment.
12. Have any infectious disease (e.g., hepatitis, tuberculosis) or a contagious immunosuppressive disease (e.g. HIV), by self-report.
13. Currently wear their contact lenes on an extended wear basis.
14. Is an employee of the investigational clinic (e.g., Investigator, Coordinator, Technician).
15. Currently wears toric or multifocal contact lenses. If the subject wears soft contact lenses for monovision, they must be willing to wear distance only correction in both eyes for the study.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 35 (Actual)
Dates: Start 2013-08; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Hong Kong Polytechnic University, Hong Hom, Kowloon, Hong Kong

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 35 subjects were enrolled in this study. Of the enrolled 1 subject did not meet the eligibility criteria.
Pre-assignment Details: Of the remaining 34 subjects, 1 subjects withdrew consent before randomization and was discontinued from the study. A total of 33 subjects were dispensed a study lens. Of the dispensed subjects 2 were discontinued and 31 completed the study. A total of 3 subjects were discontinued from this study.
Groups:
- Not Assigned: Subjects that signed the inform consent, but them withdrew consent, prior to lens dispensing.
Period: Period 1
Arm/Group | Etafilcon A/2-HEMA, EGDMA/Hefilcon A | Etafilcon A/Hefilcon A/2-HEMA, EGDMA Non-ionic | 2-HEMA, EGDMA Non-ionic/Etafilcon A/Hefilcon A | 2-HEMA, EGDMA Non-ionic/Hefilcon A/Etafilcon A | Hefilcon A/2-HEMA, EGDMA Non-ionic/Etafilcon A | Hefilcon A/Etafilcon A /2-HEMA, EGDMA Non-ionic | Not Assigned
Started | 6 | 6 | 5 | 6 | 5 | 5 | 1
Completed | 6 | 6 | 5 | 5 | 5 | 5 | 0
Not Completed | 0 | 0 | 0 | 1 | 0 | 0 | 1
Not completed — Lens Discomfort | 0 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 1
Period: Period 2
Arm/Group | Etafilcon A/2-HEMA, EGDMA/Hefilcon A | Etafilcon A/Hefilcon A/2-HEMA, EGDMA Non-ionic | 2-HEMA, EGDMA Non-ionic/Etafilcon A/Hefilcon A | 2-HEMA, EGDMA Non-ionic/Hefilcon A/Etafilcon A | Hefilcon A/2-HEMA, EGDMA Non-ionic/Etafilcon A | Hefilcon A/Etafilcon A /2-HEMA, EGDMA Non-ionic | Not Assigned
Started | 6 | 6 | 5 | 5 | 5 | 5 | 0
Completed | 6 | 6 | 5 | 5 | 4 | 5 | 0
Not Completed | 0 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Protocol Violation | 0 | 0 | 0 | 0 | 1 | 0 | 0
Period: Period 3
Arm/Group | Etafilcon A/2-HEMA, EGDMA/Hefilcon A | Etafilcon A/Hefilcon A/2-HEMA, EGDMA Non-ionic | 2-HEMA, EGDMA Non-ionic/Etafilcon A/Hefilcon A | 2-HEMA, EGDMA Non-ionic/Hefilcon A/Etafilcon A | Hefilcon A/2-HEMA, EGDMA Non-ionic/Etafilcon A | Hefilcon A/Etafilcon A /2-HEMA, EGDMA Non-ionic | Not Assigned
Started | 6 | 6 | 5 | 5 | 4 | 5 | 0
Completed | 6 | 6 | 5 | 5 | 4 | 5 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All subjects enrolled into the study.
Groups:
- Overall: All subjects that were enrolled into the study.
Arm/Group | Overall
Number analyzed (Participants) | 35
Age, Continuous [Mean (Standard Deviation); unit: Years] | 22.03 (2.885)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23
  Male | 12
Race/Ethnicity, Customized [Number; unit: Participants]
  Asian | 35
Region of Enrollment [Number; unit: Participants]
  Hong Kong | 35

OUTCOME MEASURES:

1. Primary Outcome: Corneal Staining
Description: Corneal staining was evaluated in 5 corneal regions (Central, Inferior, Nasal, Temporal and Superior) using Sodium Fluorescein strips. The corneal Staining was graded using the scale Grade 0: No Staining, Grade 1: Trace(Minimal superficial staining or stippling), Grade 2: Mild (Regional or diffuse punctate staining), Grade 3:Moderate(Significant dense coalesced staining, corneal abrasion or foreign body tracks.), Grade 4 Severe(Severe abrasions greater than 2 mm in diameter, ulcerations, epithelial loss, or full thickness abrasion.). The total was calculated by using the sum across all regions by time point. The range for the total grade for each time point would be 0-20. The total average grade for each lens and time point was evaluated as an average change from baseline level of corneal staining.
Time Frame: 20 minutes and 7 hours post lens fitting
Population: All subjects that completed every study visit without a major protocol deviation.
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: Subject Eyes
Groups:
- Etafilcon A: Subjects that received the etafilcon A lens in any of the three study periods.
- 2-HEMA, EGDMA Non-ionic: Subjects that received the 2-HEMA, EGDMA Non-ionic lens in any of the three study periods.
- Hefilcon A: Subjects that received the hefilcon A lens in any of the three study periods.
Arm/Group | Etafilcon A | 2-HEMA, EGDMA Non-ionic | Hefilcon A
Number analyzed (Participants) | 31 | 31 | 32
Number analyzed (Subject Eyes) | 62 | 62 | 64
units on a scale
  Baseline: 20 Minutes | 0.26 (0.569) | 0.15 (0.580) | 0.29 (0.624)
  7 Hours Post Lens Fitting | -0.04 (1.154) | 0.49 (1.090) | -0.02 (1.233)

ADVERSE EVENTS:
Time Frame: Throughout the duration of the study- approximately 3 days.
Arm/Group | Etafilcon A | 2-HEMA, EGDMA Non-ionic | Hefilcon A
Serious Adverse Events (participants affected / at risk) | 0/34 | 0/34 | 0/34
Other Adverse Events (participants affected / at risk) | 0/34 | 0/34 | 0/34

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days